CLINICAL TRIAL: NCT03533595
Title: Prospective Analysis of STRATAFIX Symmetric PDS Plus Suture for Fascial Closure in Spinal Surgery; Pilot Study
Brief Title: Comparative Analysis of Sutures for Fascial Closure in Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17C.580
Record Dates: First submitted 2018-04-23; First posted 2018-05-23 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Fusion of Spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Suture (No Intervention): Standard suture for thoracolumbar fusion will be used per standard of care.
- Stratafix Barbed Suture (Active Comparator): Stratafix Barbed Suture for thoracolumbar fusion will be used.
  Interventions: Device: Barbed

INTERVENTIONS:
Device: Barbed — Barbed Suture
  Arms: Stratafix Barbed Suture

SUMMARY:
STRATAFIX Symmetric PDS Plus sutures will reduce the time required for fascial closure following spinal surgery. A pilot study will aide in the design of a larger randomized controlled trial to compare suture closure time of the STRATAFIX Symmetric PDS Plus sutures versus traditional Vicryl sutures.

DETAILED DESCRIPTION:
Effective and secure suture is integral in spinal surgery, creating a strong barrier for tissue repair and a seal which prevents infection of the surgical site. The goal of any suture is to close the wound while minimizing risks of complications such as wound dehiscence and surgical site infection . A new type of suture, barbed suture, uses integrated barbs to secure the suture to the tissue without requiring knots for fixation. The result is a suture that evenly distributes tension along the length of the incision, while requiring less time to close . Additionally, STRATAFIX sutures offer a "Plus" antibacterial option for their knotless sutures, which further increases the safety and efficacy of this product.

Barbed suture technologies have been utilized in a variety of specialties, but neurosurgery remains unstudied in this respect. The primary aim of this study is to assess the time to closure using STRATAFIX technology. Decreased time to closure directly translates into decreased operating room time, and thus increased savings, especially for high-volume institutions. The secondary aim of this study is to determine the risk for surgical complications using STRATAFIX. Previous studies in other specialties have shown no significant difference in rate of adverse consequences when utilizing barbed sutures. To assess this aim, patients will be evaluated for wound dehiscence, SSI, deep infection, and 30-day rate of readmission for wound infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old
2. Patients undergoing thoracolumbar fusion of at least 3 vertebral levels.
3. Patient able to sign informed consent.

Exclusion Criteria:

1. Current infection (osteomyelitis), diabetes, severely malnourished or other co-morbidities that the investigator believes does not make the patient a good candidate for surgery.
2. Patients with incidental durotomy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Reduced operating times | Patient followed for 6 months from surgery
  STRATAFIX Symmetric PDS Plus sutures will reduce the time required for fascial closure following spinal surgery. A pilot study will aide in the design of a larger randomized controlled trial to compare suture closure time of the STRATAFIX Symmetric PDS Plus sutures versus traditional Vicryl sutures.

SECONDARY OUTCOMES:
Safety evaluation of wound dehiscence | Patient followed for 6 months from surgery
  Subject's surgical site wound will be monitored during the protocol defined time points.
Safety evaluation of surgical site infection (SSI) rate | Patient followed for 6 months from surgery
  Subject's surgical site will be monitored and assessed for infection during the protocol defined time points.
Safety evaluation of 30 days readmission rates | Patient followed for 30 days from surgery
  Subject will be monitored for 30 days post surgery for AE's and SAE's which result in readmission to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Heller, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided